CLINICAL TRIAL: NCT07167745
Title: SMALL BOWEL INCIDENTAL STRICTURES: EVALUATION OF NATURAL HISTORY IN ASYMPTOMATIC CROHN'S EVOLUTION (SILENCE STUDY)
Brief Title: Tracking the Natural Course of Silent Small Bowel Narrowing in Adults With Crohn's Disease
Acronym: SILENCE
Status: Completed | Type: Observational
Sponsor: University Medical Center Zvezdara (Other)
Collaborators: Centre Hospitalo-Universitaire de Brabois, Vandoeuvre Les Nancy, France (Unknown)
Responsible Party: Principal Investigator, Tamara Knezevic Ivanovski, Teaching assistent, University Medical Center Zvezdara
Other Study IDs: IRB00009457, IORG0007877; IRB00009457, IORG0007877 (Other: University Hospital Zvezdara)
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Incidentally Diagnosed Asymptomatic Small Bowel Strictures at Crohn's Disease Diagnosis: Adults (≥18 years) with Crohn's disease whose asymptomatic small bowel stricture was discovered at the same time as their initial Crohn's disease diagnosis. All were in clinical remission at baseline and had no gastrointestinal symptoms related to obstruction. Strictures were confirmed by MR enterography, intestinal ultrasound, or endoscopy. Follow-up data were collected retrospectively for at least 12 months to evaluate progression to symptoms, changes in stricture morphology, and need for medical, endoscopic, or surgical intervention.

SUMMARY:
Crohn's disease is a long-term condition that causes inflammation in the digestive tract. Over time, some people develop narrowings in the small intestine, called "strictures." These strictures can block food and cause symptoms like abdominal pain, bloating, nausea, or vomiting. However, strictures are sometimes found by chance in people who have no symptoms. These are called "asymptomatic" or "silent" strictures.

Doctors do not know how often silent strictures become a problem or whether it is better to treat them early or simply monitor them. Current treatments for Crohn's disease are not very effective at reversing scar tissue once it forms, and there are no clear guidelines for what to do when a silent stricture is found.

The SILENCE study will look at the natural course of silent small bowel strictures in adults with Crohn's disease. Researchers will review the medical records of people aged 18 and older who were diagnosed with a silent small bowel stricture between 2015 and 2023. All participants must have at least one year of follow-up information available.

The study will record:

How often strictures become symptomatic (cause abdominal pain, nausea, vomiting, bloating, or other symptoms)

Whether patients require treatments such as changes in medication, endoscopic dilation, or surgery

Any changes in the size or severity of the stricture seen on imaging or endoscopy

The study will also compare two groups:

People whose silent stricture was found at the same time as their Crohn's diagnosis

People with Crohn's in remission for at least two years before developing a silent stricture

Researchers will examine possible risk factors for progression, such as age, smoking status, prior treatment, and results from blood or stool tests.

By understanding how silent strictures behave over time, this study aims to help doctors decide when it is safe to observe and when intervention might be needed. The findings could improve patient care and inform future treatment guidelines for Crohn's disease.

DETAILED DESCRIPTION:
SMALL BOWEL INCIDENTAL STRICTURES: EVALUATION OF NATURAL HISTORY IN ASYMPTOMATIC CROHN'S EVOLUTION (SILENCE STUDY)

Crohn's disease (CD) is a progressive, chronic inflammatory disorder of the gastrointestinal tract, classically categorized into three phenotypes: inflammatory, stricturing, and penetrating (1). While most patients initially present with the inflammatory phenotype, the disease can evolve over time into stricturing or penetrating forms due to recurrent cycles of inflammation leading to cumulative bowel damage (2). Typically, CD is diagnosed following the onset of gastrointestinal symptoms and subsequent endoscopic evaluation. However, a subset of patients may be incidentally diagnosed with CD, including small bowel strictures, during imaging or colonoscopy performed for unrelated indications(3). Although the most common cause is CD, strictures in the small bowel also may result from various etiologies, such as prior surgery, radiation enteritis, NSAID-induced injury, or congenital anomalies.

Among patients with CD, the terminal ileum is the most frequently involved site of stricturing disease. While approximately 10% of patients initially present with a stricturing phenotype, the risk of developing strictures increases over time estimated at 15% by 10 years and over 20% by 20 years after diagnosis(4). Importantly, 40-70% of patients with fibrostenotic CD will eventually require surgical intervention due to complications such as obstruction or failure of medical therapy(5). Nevertheless, not all strictures cause symptoms immediately - an estimated ~17% of small-bowel CD may be asymptomatic when detected (6). Despite the availability of advanced medical therapies, current treatment options have shown limited effectiveness in preventing or reversing intestinal strictures in CD(7-9). Much of the current epidemiologic data is derived from the Vienna and Montreal classification systems, which are based primarily on symptomatic disease(5). As such, the true burden of asymptomatic fibrostenotic CD may be underrecognized. Small bowel strictures may be incidentally detected in asymptomatic patients undergoing imaging or endoscopy for unrelated reasons, raising important clinical questions regarding their natural history and optimal management. The optimal management of incidentally found, asymptomatic strictures remain unclear; there are currently no firm guidelines on whether to intervene early or simply observe. For example, no clear consensus exists on managing an incidental stricture in an asymptomatic patient - endoscopic dilation might delay progression, but any proactive intervention must balance potential benefits against risks(4,6,10). Consequently, despite the widespread use of biologics, the incidence of strictures in CD has remained largely unchanged.

Pathogenesis of Fibrosis Stricture formation is a slow process and only becomes apparent in late stages, which is why antecedent events are hard to study. It is a dynamic process where mediators, cell populations, and physical conditions change over time; it is also intuitive to think that stricture location (ileum vs colon) likely matters(11). The development of intestinal fibrosis involves a complex interplay between inflammation-dependent and inflammation-independent mechanisms. A key feature is the persistent activation of mesenchymal cells, leading to excessive deposition of extracellular matrix (ECM) components. Fibrosis leads to thickening of all intestinal wall layers, including mucosa and muscularis mucosa, submucosa which is often filled with dense collagen bands (predominantly collagen types III and V and fibronectin and tenascin C) and smooth muscle cell islands, muscularis propria(12,13). Natural history, how these lesions progress over time, is not well documented. It is widely assumed that once a stricture forms it will gradually worsen, yet robust longitudinal data confirming this progressive behavior are lacking(14).

Clinical Implications Even in the absence of symptoms, asymptomatic strictures may represent subclinical disease progression and pose risks for future bowel obstruction, bacterial overgrowth, or complications requiring intervention. Current medical therapies have limited ability to reverse or prevent fibrotic changes, highlighting the need for early detection, monitoring, and research into antifibrotic strategies. A comprehensive review of the literature revealed that no studies to date have specifically addressed asymptomatic small bowel strictures in CD and their natural history. However, a limited number of studies have included small cohorts of patients diagnosed with asymptomatic CD including asymptomatic strictures (3,10,15). Those studies indicated that these remained largely symptom-less and without apparent disease progression throughout several years of follow-up despite receiving no specific treatment (3,10). However, considering the small number of patients and the fact that asymptomatic strictures wer

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are asymptomatic, with no clinical signs of intestinal symptomatology (absence of abdominal pain, distension, nausea, vomiting, weight loss, diahorrea).

  * Patients 18 years and older
  * Small bowel stricture diagnosed incidentally either:

    1. at the time of initial Crohn's disease (CD) diagnosis (baseline visit), or
    2. in patients with a previously established diagnosis of mild CD who have maintained stable clinical, endoscopic and radiographic remission without previous stenosis for a minimum of 2 years prior to study entry.
  * Diagnosis of Crohn's disease confirmed according to accepted clinical, endoscopic, radiologic, and/or histologic standards.
  * Evidence of small bowel involvement by CD, either in the form of ileal, ileocolonic or jejunal disease. Presence of a small bowel stricture confirmed by MR enterography, intestinal ultrasound (IUS), or endoscopy.
  * Only patients who have at least one year of longitudinal follow-up data in the medical record after the baseline/index evaluation will be included.
  * Patients who went to colonoscopy due to asymptomatic iron deficiency anemia and/or positive fecal occult blood test or for routine CD follow up
  * Minimum follow up period is one year, or event happened whichever comes first

Exclusion Criteria:

* Presence of symptomatic strictures at the time of stenosis detection.
* Incomplete clinical data or follow-up
* Strictures attributable to neoplastic processes, prior radiation therapy, or congenital anomalies.
* Strictures are located exclusively in the colon.
* Clinical symptoms of active CD at the time the stricture was identified.
* History of prior small bowel or colonic resection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective multicenter study will include patients aged above 18 years diagnosed with asymptomatic small bowel strictures between 2015 and 2023, with a minimum follow-up of one year, selected based on predefined inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Proportion of asymptomatic small bowel strictures in Crohn's disease patients that progress to symptomatic disease | From baseline to last available follow-up, minimum 12 months, up to 5 years
  Percentage of patients with incidentally detected, asymptomatic small bowel strictures who develop symptoms consistent with sub-obstruction (abdominal pain, nausea, vomiting, bloating) during the follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zvezdara, Belgrade, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the findings of this study will be shared. This includes baseline demographics, clinical characteristics, imaging and endoscopic findings, laboratory results, treatment details, and outcomes related to the progression of asymptomatic small bowel strictures in Crohn's disease. All personal identifiers will be removed to protect participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available starting 6 months after publication of the primary results and will remain available for 5 years.
Access Criteria: Data will be made available to qualified researchers whose proposed use of the data has been reviewed and approved by the study steering committee. Proposals should include a research plan and justification for data use.